CLINICAL TRIAL: NCT02164526
Title: National, Prospective, Multicenter,Observational Registry Study on Pulmonary Hypertension Due to Left Heart Disease in China
Brief Title: Registry for Pulmonary Hypertension Due to Left Heart Disease in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Director of Pulmonary vascular disease center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CRPHDLHD
Record Dates: First submitted 2014-06-04; First posted 2014-06-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Hypertension Due to Left Heart Disease
Keywords: Pulmonary Hypertension; Left Heart Disease; Heart failure; Registry; China
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment
  Interventions: Other: Routine therapy

INTERVENTIONS:
Other: Routine therapy — Routine therapy

SUMMARY:
Left heart disease is the main cause of pulmonary hypertension. With the advent of the aging society, chronic heart failure has become a global public health problem. Therefore the prevalence of pulmonary hypertension due to the left heart disease is increasing. However, there is no research on the prevalence of pulmonary hypertension due to the left heart disease in China. Therefore, the aim of the present study was to describe real-world outcome of Chinese patients with pulmonary hypertension due to the left heart disease and identify factors that may predict outcome. Our study will profile the demographics, clinical course, treatments, and outcomes of pulmonary hypertension due to the left heart disease in China.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Hypertension due to left heart disease

Exclusion Criteria:

* Other forms of Pulmonary Hypertension
* Heart failure due to valvular heart disease
* Hypertrophic obstructive cardiomyopathy
* Right ventricular outflow tract stenosis
* Pericardial disease
* Patients with chronic lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who were diagnosed as pulmonary hypertension due to the left heart disease in 35 participating institutions in China
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
All cause death | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Huang L, Pang L, Gu Q, Yang T, Li W, Quan R, Su W, Wu W, Tang F, Zhu X, Shen J, Sun J, Shan G, Xiong C, Huang S, He J. Prevalence, risk factors, and survival associated with pulmonary hypertension and heart failure among patients with underlying coronary artery disease: a national prospective, multicenter registry study in China. Chin Med J (Engl). 2022 Aug 5;135(15):1837-1845. doi: 10.1097/CM9.0000000000002112. PMID 36195993
- [Derived] Lin Y, Pang L, Huang S, Shen J, Wu W, Tang F, Su W, Zhu X, Sun J, Quan R, Yang T, Han H, He J. Impact of borderline pulmonary hypertension due to left heart failure on mortality in a multicenter registry study: A 3-year survivorship analysis. Front Cardiovasc Med. 2022 Aug 12;9:983803. doi: 10.3389/fcvm.2022.983803. eCollection 2022. PMID 36035936
- [Derived] Quan R, Huang S, Pang L, Shen J, Wu W, Tang F, Zhu X, Su W, Sun J, Yu Z, Wang L, Zhu X, Xiong C, He J. Risk prediction in pulmonary hypertension due to chronic heart failure: incremental prognostic value of pulmonary hemodynamics. BMC Cardiovasc Disord. 2022 Feb 16;22(1):56. doi: 10.1186/s12872-022-02492-1. PMID 35172722